CLINICAL TRIAL: NCT05549934
Title: A Pilot Study to Assess Safety and Biomarker Responses of Ritlecitinib (JAK3/TEC Inhibitor) in Cicatricial Alopecia
Brief Title: Ritlecitinib for Cicatricial Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emma Guttman (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Emma Guttman, The Waldman Professor and System Chair, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 22-1234
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cicatricial Alopecia
Keywords: frontal fibrosing alopecia; FFA; lichen planopilaris; LPP; central centrifugal; scarring alopecia; CCCA
MeSH Terms: conditions — Alopecia; Lichen Planus | interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06651600 (Ritlecitinib) (Experimental): 200 mg once-daily for 8 weeks and then 100 mg once daily for the remaining 40 weeks
  Interventions: Drug: PF-06651600

INTERVENTIONS:
Drug: PF-06651600 — tablets containing active drug (a combined JAK3/TEC inhibitor)
  Other Names: Ritlecitinib

SUMMARY:
Alopecia could be subdivided into two main groups of diseases: non-scarring alopecia, such as male pattern baldness, or alopecia areata (AA), in which hair follicles are preserved, yet quiescent, and scarring alopecia, also known as cicatricial alopecia (CA), in which hair follicles are irreversibly destroyed. CA leads to scarred areas, most commonly on the scalp, that cannot re-grow hair. Despite being a long-term condition, that often has significant impact on patients' well-being, available effective treatments for these diseases are lacking. In addition, the molecular abnormalities causing CA are largely unknown. The research team will be administering a new investigational drug (a JAK3/TEC inhibitor), ritlecitinib, which has shown statistically significant improvement in scalp hair loss for AA patients in a proof of concept and phase 2b/3 studies (B7981015 AA study). This is an open-label clinical trial. CA patients will be asked to provide small samples of skin and blood throughout the treatment period, to find out how they respond to the drug, and to attempt to better understand these diseases.

ELIGIBILITY:
INCLUSION CRITERIA

* Subjects of any gender, age 18 years or older, at the time of informed consent at Screening
* Subjects who are willing and able to adhere to the study visit schedule and comply with protocol requirements.
* Subject self-reports a history of at least 6 months of CA (LPP/FFA or CCCA). Diagnosis will be made clinically (according to the LPPAI37, FFASI36 and/or CHLG38).
* Subject has a negative Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) at screening or within the last 12 months.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) OR;
  * Is a WOCBP (all female participants, regardless of whether or not they have experienced/reported menarche, are considered WOCBP unless they are permanently sterile or confirmed infertile). A WOCBP who is sexually active must use a contraceptive method that is highly effective, with a failure rate of <1%, during the intervention period and for at least 28 days after the last dose of study intervention.
  * And if a WOCBP, must have a negative highly sensitive serum pregnancy test at the screening visit and a negative urine pregnancy test at baseline performed before the first dose of study intervention.
* Subject is judged to be in otherwise good overall health following a detailed medical and medication history, physical examination, and laboratory testing.

EXCLUSION CRITERIA

* Subject's cause of hair loss is indeterminable and/or they have concomitant causes of alopecia, such pregnancy-related, drug-induced, telogen effluvium, or advanced androgenetic alopecia.
* Subject has a history of CA for ≥ 7 years since their disease onset, severe fibrosing disease, or very rapid hair loss at screening (de novo patients only).
* Subject has a history of moderate to severe keloids on the scalp, as determined by clinical examination at screening.
* Other scalp disease that may impact assessment (e.g., scalp psoriasis, dermatitis, etc.).
* Subject is pregnant or breastfeeding.
* Participation in other studies involving investigational drug(s) within 4 weeks or within 5 half-lives (if known), whichever is longer, prior to study entry and/or during study participation (de novo patients only).
* Active systemic diseases that may cause hair loss (e.g., systemic lupus erythematosus, thyroiditis, systemic sclerosis, etc.).
* Any Psychiatric condition in the opinion of the investigator precludes participation in the study.
* Subjects with a Columbia Suicide Severity Rating Scale (C-SSRS) score of "yes" on questions 4 and/or 5 at Visit 2 (Baseline).
* Current or recent history of clinically significant severe, progressive, or uncontrolled renal (including but not limited to active renal disease or recent kidney stones), hepatic, hematological, gastrointestinal, metabolic, endocrine (particularly thyroid disease which can be associated with hair loss), pulmonary, cardiovascular, psychiatric, immunologic/rheumatologic or neurologic disease; or have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or interfere with the interpretation of study results; or in the opinion of the investigator, the subject is inappropriate for entry into this study, or unwilling/unable to comply with STUDY PROCEDURES.
* History of thromboembolic events including DVT and PE or history of inherited coagulopathies.
* Any present malignancies or history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* History of any lymphoproliferative disorder such as Epstein Barr Virus (EBV) related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
* History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
* History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 0.
* Active acute or chronic infection requiring treatment with oral antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to Day 0 or superficial skin infection within 1 week prior to Day 0.
* Significant trauma or major surgery within 1 month of signing informed consent.
* Considered in imminent need for surgery or with elective surgery scheduled to occur during the study.
* Active hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or positive HIV serology at the time of screening for subjects determined by the investigators to be at high-risk for this disease.
* ANY of the following abnormalities in the clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary:

  * Absolute neutrophil count of <1.2 x 109/L (<1200/mm3);
  * Hemoglobin <11.0 g/dL or hematocrit <33%;
  * Platelet count of <150 x 109/L (<150,000/mm3);
  * Absolute lymphocyte count of <0.80 x 109 /L (<800/mm3);
  * Estimated Glomerular Filtration Rate (eGFR) less than 60 mL/ml/min/1.73m2 based on CKD-Epi 2021 (creatine equation);
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values >2 times the ULN;
  * Total bilirubin greater than or equal to 1.5 times the ULN; participants with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is less than or equal to ULN.
* Have an active history of alcohol or substance abuse within 1 year prior to Day 0.
* Donation of blood in excess of 500 mL within 8 weeks prior to Day 0.
* Subject has received a live attenuated vaccine ≤ 6 weeks prior to study screening.
* Subject has any uncertain or clinically significant laboratory abnormalities that may affect interpretation of study data or endpoints, at determined by the PI.
* History of adverse systemic or allergic reactions to components of study drug.
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, within 8 weeks prior to baseline visit.
* Use of other non-biologic systemic agent for CA, including, 5α-reductase inhibitors, hydroxychloroquine, or retinoids, within 4 weeks prior to baseline visit.
* Use of an intralesional corticosteroids or oral JAK inhibitor (tofacitinib, ruxolitinib, or any JAK1/TYK2 product) within 4 weeks prior to the baseline visit (de novo patients only).
* Subject has used topical corticosteroids, and/or tacrolimus, and/or pimecrolimus or cyclosporine within 1 week before the baseline visit.
* Subject has been previously treated with biological drugs in the last 12 weeks for other indications.
* Subjects previously tested with a positive or indeterminable PPD or QFT result, including subjects that completed standard tuberculosis therapy.
* Screening 12-lead ECG that demonstrates clinically significant abnormalities requiring treatment, e.g. acute myocardial infarction, serious tachy or brady arrhythmias or that are indicative of serious underlying heart disease (e.g. cardiomyopathy, major congenital heart disease, low voltage in all leads, Wolff-Parkinson-White syndrome and other clinically relevant abnormalities which may affect participant safety or interpretation of study results. A history of additional risk factors for Torsades de Pointes (TdP) (e.g. heart failure, hypokalemia, family history of long QT syndrome).
* If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated 2 more times and the average of 3 QTc or QRS values should be used to determine the participants' eligibility. Participants with average screening value QTcF > 450 ms should be excluded.
* The use of prohibited and permitted CYP3A substrates are provided in Appendix 2.1 and 2.2, respectively and medications that prolong the QT/QTcF interval in Appendix 3.
* Have hearing loss with progression over the previous 5 years, or sudden hearing loss, or middle or inner ear disease such as otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered acute, fluctuating, or progressive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events | Week 48
  The adverse event will be described and categorized as Treatment-emergent, Serious, abnormal in vital signals, and abnormalities in laboratory parameters.
Severity of Treatment-Emergent Adverse Events | Week 48
  The adverse event will be categorized according to CTCAE guidelines when applicable
Change in Ct values of mRNA levels of CCL5 gene | Baseline to Week 24
  Changes in mRNA Levels of CCL5 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline and week 24. The unit of the outcome is called Ct value and it represents the number of amplification cycles to reach a level of fluorescence in the experiment. The Ct value is directly associated to the level of expression of a gene
Change in Ct values of mRNA levels of CCL5 gene | Baseline to Week 48
  Changes in mRNA Levels of CCL5 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline and week 48. The unit of the outcome is called Ct value and it represents the number of amplification cycles to reach a level of fluorescence in the experiment. The Ct value is directly associated to the level of expression of a gene.

SECONDARY OUTCOMES:
Change in Ct values of mRNA levels of CXCR3 | Baseline to Week 24
  Changes in mRNA Levels of CXCR3 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline and week 24. The unit of the outcome is called Ct value and it represents the number of amplification cycles to reach a level of fluorescence in the experiment. The Ct value is directly associated to the level of expression of a gene.
Ct value of mRNA levels of CXCR3 | Baseline to Week 48
  Changes in mRNA Levels of CXCR3 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline and week 48. The unit of the outcome is called Ct value and it represents the number of amplification cycles to reach a level of fluorescence in the experiment. The Ct value is directly associated to the level of expression of a gene.
The Frontal Fibrosis Alopecia Severity Index (FFASI) | Baseline
  The Frontal Fibrosis Alopecia Severity Index utilizes clinical images of the entire hairline from a total score of 0-84, with higher score indicating more severity.
The Frontal Fibrosis Alopecia Severity Index (FFASI) | Week 24
  The Frontal Fibrosis Alopecia Severity Index utilizes clinical images of the entire hairline, from a total score of 0-84, with higher score indicating more severity.
The Frontal Fibrosis Alopecia Severity Index (FFASI) | Week 48
  The Frontal Fibrosis Alopecia Severity Index utilizes clinical images of the entire hairline, from a total score of 0-84, with higher score indicating more severity.
The Lichen Planopilaris Activity Index (LPPAI) | Baseline
  The Lichen Planopilaris Activity Index is a numeric composite index that aggregates symptoms and signs of pruritus, pain, burning, scalp erythema , perifollicular erythema, perifollicular scale , pull test and spreading. Symptoms and signs are measured in a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe). Full range from 0-10, higher score indicates more severity.
The Lichen Planopilaris Activity Index (LPPAI) | Week 24
  The Lichen Planopilaris Activity Index is a numeric composite index that aggregates symptoms and signs of pruritus, pain, burning, scalp erythema , perifollicular erythema, perifollicular scale , pull test and spreading. Symptoms and signs are measured in a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe). Full range from 0-10, higher score indicates more severity.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman-Yassky, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Not shared

DOCUMENTS (1):
  • Informed Consent Form (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT05549934/ICF_001.pdf